CLINICAL TRIAL: NCT02097030
Title: Single-Center Clinical Evaluation of Daily Disposable Contact Lenses
Brief Title: Clinical Evaluation of Daily Disposable Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: EX-MKTG-46
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- etafilcon A lens (Active Comparator): Participants were randomized to either the etafilcon A or the nelfilcon A lens for three days and then both groups wore the filcon II 3 lens for three days, without washout period between lens types.
  Interventions: Device: etafilcon A
- nelfilcon A lens (Active Comparator): Participants were randomized to either the etafilcon A or the nelfilcon A lens for three days and then both groups wore the filcon II 3 lens for three days, without washout period between lens types.
  Interventions: Device: nelfilcon A
- filcon II 3 lens (Active Comparator): Participants were randomized to either the etafilcon A or the nelfilcon A lens for three days and then both groups wore the filcon II 3 lens for three days, without washout period between lens types.
  Interventions: Device: filcon II 3

INTERVENTIONS:
Device: filcon II 3 — Participants wear a first pair of lenses for three days and then crossover and wear a second pair of lenses for three days.
  Other Names: Silicone Hydrogel Daily Disposable Contact Lens
  Arms: filcon II 3 lens
Device: etafilcon A — Participants wear a first pair of lenses for three days and then crossover and wear a second pair of lenses for three days.
  Other Names: Hydrogel Daily Disposable Contact Lens
  Arms: etafilcon A lens
Device: nelfilcon A — Participants wear a first pair of lenses for three days and then crossover and wear a second pair of lenses for three days.
  Other Names: Hydrogel Daily Disposable Contact Lens
  Arms: nelfilcon A lens

SUMMARY:
The objective of the study is to compare the overall subjective preference of filcon II 3 daily disposable silicone hyrogel contact lenses compared to etafilcon A and nelfilcon A daily disposable conventional hydrogel contact lenses.

DETAILED DESCRIPTION:
Double-masked, randomised, controlled crossover trial. Subjects were randomized to wear one or the other of the conventional hydriogel lenses; all subjects wore the filcon II 3 lenses. The first randomly assigned lens type was worn for 3 days, with daily replacement, followed by 3 days of wear of the other lens type, with daily replacement.

ELIGIBILITY:
Inclusion Criteria:

* Is between 18 and 40 years of age (inclusive)
* Has had a self-reported visual exam in the last two years
* Is an adapted soft CL wearer
* Must be able to wear their lenses at least 3 full days, 10 hours per day, assuming there are no contraindications for doing so
* Has a CL spherical prescription between - 1.00 and - 6.00 (inclusive)
* Has less than 1.25 D spectacle cylinder in each eye.
* Baseline vision of 20/40 or better (in each eye) with their habitual vision correction or 20/20 best-corrected.
* Is correctable to at least 20/25 distance visual acuity with study contact lenses in each eye
* Has clear corneas and no active ocular disease
* Has read, understood and signed the information consent letter
* Is willing to comply with the wear schedule (at least 3 full days)
* Is willing to comply with the visit schedule

Exclusion Criteria:

* Has never worn contact lenses before.
* Currently wears rigid gas permeable contact lenses.
* Has a history of not achieving comfortable CL wear (3 days per week; > 8 hours/day)
* Has a CL prescription outside the range of - 1.00 to -6.00D
* Has a spectacle cylinder greater than -1.25D of cylinder in either eye.
* Has best corrected spectacle distance vision worse then 20/25 in either eye.
* Has any systemic disease affecting ocular health.
* Is using any systemic or topical medications, (includes rewetting drops, artificial tears and allergy drops), that will affect ocular health. Occasional use is acceptable but not during the trial.
* Has any ocular pathology or severe insufficiency of lacrimal secretion
* Has persistent, clinically significant corneal or conjunctival staining
* Has active neovascularization or any central corneal scars.
* Is aphakic.
* Is presbyopic.
* Has undergone corneal refractive surgery.
* Is participating in any other type of eye related clinical or research study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2014-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng C Lin, OD, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley Clinical Research Center (UCB-CRC), Berkeley, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single center evaluation. Thirty five subjects were recruited and 30 subjects completed the trial.
Pre-assignment Details: Three participants were enrolled in the study but did not meet inclusion criteria, therefore discontinued before lens randomization.
Groups:
- Etafilcon A, Then Filcon II 3: Participants wear a first pair of lenses for three days and then crossover and wear a second pair of lenses for three days.
  etafilcon A: contact lens filcon II 3: contact lens
- Nelfilcon A, Then Filcon II 3: Participants wear a first pair of lenses for three days and then crossover and wear a second pair of lenses for three days.
  nelfilcon A: contact lens filcon II 3: contact lens
Period: First Intervention (3 Days)
Arm/Group | Etafilcon A, Then Filcon II 3 | Nelfilcon A, Then Filcon II 3
Started | 15 | 17
Completed | 14 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Visual Acuity | 0 | 1
Period: Second Intervention (3 Days)
Arm/Group | Etafilcon A, Then Filcon II 3 | Nelfilcon A, Then Filcon II 3
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etafilcon A, Then Filcon II 3 | Nelfilcon A, Then Filcon II 3 | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (4.9) | 21.2 (5.0) | 21.4 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Lens Preference - All Study Lenses
Description: Participant's subjective response for overall lens preference after 3 days of daily disposable wear of each pair of lenses. Surveyed at exit. (4 possible ratings: Strongly prefer pair#1, Slightly prefer pair #1, Slightly prefer pair #2, Strongly prefer pair #2).
Time Frame: Study Exit
Population: Subjects were randomized to wear one or the other of the conventional hydrogel lenses; all subjects wore the Clariti silicone hydrogel lenses.
Measure: Number; unit: participants
Groups:
- Nelfilcon A; Etafilcon A; Filcon II 3: Subjects randomized to wear study pair one then crossover to study pair two. Study pairs are either filcon II 3 and nelfilcon A or filcon II 3 and etafilcon A
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Strongly Prefer | 5 | 3 | 8
  Slightly Prefer | 4 | 3 | 7

2. Primary Outcome: Overall Lens Preference - Hydrogel vs. Filcon II 3
Description: Participant's subjective response for overall lens preference after 3 days of daily disposable wear of each pair. Surveyed at exit. (4 possible ratings: Strongly prefer pair#1, Slightly prefer pair #1, Slightly prefer pair #2, Strongly prefer pair #2).
Time Frame: Study Exit
Population: 30 subjects
Measure: Number; unit: participants
Groups:
- Hydrogel; Filcon II 3: Subjects randomized to wear study pair one then crossover to study pair two. Study pairs are either filcon II 3 and nelfilcon A or filcon II 3 and etafilcon A.
  (hydrogel: nelfilcon A, etafilcon A) (silicone hydrogel: filcon II 3)
Arm/Group | Hydrogel | Filcon II 3
Number analyzed (Participants) | 30 | 30
participants
  Strongly Prefer | 8 | 8
  Slightly Prefer | 7 | 7

3. Secondary Outcome: Subjective Response for Comfort
Description: Participant's subjective response for comfort measured at baseline and 3 day follow-up. (Continuous Comfort Scale 0-100, 0=cannot be worn/causes pain, 100=cannot be felt ever)
Time Frame: Baseline and 3 day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 90.3 (15.9) | 94.1 (8.7) | 93.2 (9.5)
  3 day follow up | 84.5 (12.2) | 82.0 (16.3) | 81.5 (20.1)

4. Secondary Outcome: Subjective Response for Vision
Description: Participant's subjective response for vision measured at baseline and at 3 day follow-up of daily disposable wear of lenses. (Vision Scale 0-100, 0=very blurry, 100=very clear).
Time Frame: Baseline and 3 day follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 93.8 (8.2) | 93.0 (9.6) | 94.1 (6.1)
  3 day follow up | 94.8 (5.4) | 90.6 (15.8) | 95.2 (5.1)

5. Secondary Outcome: Subjective Response for Insertion
Description: Participant's subjective response for insertion measured at baseline. (Insertion Handling Scale 0-100, 0=very hard to handle, 100=very easy to handle).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale | 94.6 (8.5) | 86.4 (18.4) | 91.0 (15.1)

6. Secondary Outcome: Subjective Response for Handling (Insertion and Removal)
Description: Participant's subjective response for handling (insertion and removal) measured at 3 day follow-up of daily disposable wear of lenses. (Handling Scale 0-100, 0=very hard to handle, 100=very easy to handle).
Time Frame: 3 days follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Insertion | 92.9 (11.6) | 74.1 (23.6) | 91.3 (10.1)
  Removal | 88.6 (14.8) | 94.8 (8.0) | 93.9 (11.8)

7. Secondary Outcome: Subjective Response for Dryness
Description: Participant's subjective response for dryness, measured at baseline and after 3 day follow-up of daily disposable wear of lenses. (Dryness Scale 0-100, 0=Cannot be worn/extremely dry, 100=no dryness experienced at any time).
Time Frame: 3 Days Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale | 80.6 (16.8) | 81.6 (19.0) | 76.4 (21.5)

8. Secondary Outcome: Overall Satisfaction, Vision
Description: Participant's subjective response for overall vision satisfaction. Measured after 3 days daily disposable wear of lenses. (4 point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied.
Time Frame: 3 Days Follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Completely Dissatisfied | 0 | 0 | 0
  Somewhat Dissatisfied | 0 | 1 | 0
  Somewhat Satisfied | 2 | 2 | 6
  Completely Satisfied | 14 | 11 | 24

9. Secondary Outcome: Overall Satisfaction, Comfort
Description: Participant's subjective response for overall comfort satisfaction. Measured after 3 days daily disposable wear of lenses. (4 point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied.
Time Frame: 3 Days Follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Completely Dissatisfied | 0 | 0 | 0
  Somewhat Dissatisfied | 3 | 1 | 5
  Somewhat Satisfied | 5 | 8 | 9
  Completely Satisfied | 8 | 5 | 16

10. Secondary Outcome: Overall Satisfaction, Handling
Description: Participant's subjective response for overall handling satisfaction. Measured after 3 days of daily disposable lens wear. (4 point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied.
Time Frame: 3 Days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Completely Dissatisfied | 0 | 0 | 0
  Somewhat Dissatisfied | 1 | 4 | 4
  Somewhat Satisfied | 6 | 3 | 10
  Completely Satisfied | 9 | 7 | 16

11. Secondary Outcome: Overall Satisfaction, Dryness
Description: Participant's subjective response for overall dryness satisfaction. Measured after 3 days daily disposable wear of lenses. (4 point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied.
Time Frame: 3 Days Follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Completely Dissatisfied | 1 | 0 | 2
  Somewhat Dissatisfied | 4 | 3 | 5
  Somewhat Satisfied | 6 | 5 | 12
  Completely Satisfied | 5 | 6 | 11

12. Secondary Outcome: Overall Satisfaction
Description: Participant's subjective response for overall satisfaction. Measured after 3 days of daily disposable lens wear. (4 point Likert Scale; Completely Satisfied, Somewhat Satisfied, Somewhat Dissatisfied, Completely Dissatisfied.
Time Frame: 3 Days Follow-up
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
participants
  Completely Dissatisfied | 0 | 0 | 1
  Somewhat Dissatisfied | 1 | 1 | 3
  Somewhat Satisfied | 8 | 9 | 11
  Completely Satisfied | 7 | 4 | 15

13. Secondary Outcome: Lens Fit and Performance - Wettability (Baseline and 3 Days Follow-up)
Description: The investigator's objective assessment for contact lens fit and performance - wettability. Measured at baseline (10-15mins settling) for both study pairs. Wettability (scale 0-4, 0.25 steps, 0=excellent, 4 severely reduced).
Time Frame: Baseline and 3 days follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 3.5 (0.3) | 3.3 (0.5) | 3.4 (0.4)
  3 days follow up | 3.6 (0.2) | 3.2 (0.6) | 3.5 (0.4)

14. Secondary Outcome: Lens Fit and Performance - Deposits (Baseline and 3 Days Follow-up)
Description: The investigator's objective assessment for contact lens fit and performance - deposits. Measured at baseline (10-15mins settling) for both study pairs. Deposits (scale 0-4, 0.25 steps, 0=excellent, 4 severely reduced);
Time Frame: Baseline and 3 days follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 0.0 (0.0) | 0.1 (0.3) | 0.0 (0.0)
  3 days follow up | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)

15. Secondary Outcome: Lens Fit and Performance - Debris (Baseline and 3 Day Follow-up)
Description: The investigator's objective assessment for contact lens fit and performance - debris. Measured at baseline (10-15mins settling) for both study pairs. (Debris scale 0-4; 0.25 steps; 0=no debris, 4=significant debris)
Time Frame: Baseline and 3 day follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 0.0 (0.0) | 0.0 (0.0) | 0.0 (0.0)
  3 days follow up | 0.0 (0.0) | 0.0 (0.0) | 0.1 (0.6)

16. Secondary Outcome: Lens Fit and Performance - Movement (Baseline and 3 Days Follow-up)
Description: The investigator's objective assessment for contact lens fit and performance - movement. Measured at baseline (10-15mins settling) for both study pairs. Movement (scale in millimeters).
Time Frame: Baseline and 3 days follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 0.3 (0.2) | 0.3 (0.2) | 0.3 (0.1)
  3 days follow up | 0.2 (0.2) | 0.3 (0.2) | 0.3 (0.2)

17. Secondary Outcome: Lens Fit and Performance - Fit Acceptance
Description: The investigator's objective assessment for contact lens fit and performance - fit acceptance. Measured at baseline and 3 day follow-up (10-15mins settling) for both study pairs. Fit acceptance (Scale 0-4, 0.25 steps, 0=Should not be worn, 4=Perfect).
Time Frame: Baseline and 3 day follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 3.6 (0.2) | 3.6 (0.2) | 3.7 (0.2)
  3 days follow up | 3.6 (0.3) | 3.6 (0.2) | 3.7 (0.2)

18. Secondary Outcome: Lens Fit and Performance - Tightness (Baseline and 3 Day Follow-up)
Description: The investigator's objective assessment for contact lens fit and performance - tightness. Measured at baseline (10-15mins settling) for both study pairs. Tightness (Scale 0-4, 0.25 steps, 0=Should not be worn, 4=Perfect).
Time Frame: Baseline and 3 day follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Baseline | 54.0 (12.0) | 56.0 (11.0) | 53.0 (12)
  3 days follow up | 58.0 (12) | 55 (12.0) | 54 (11)

19. Secondary Outcome: Ocular Health - Biomicroscopy
Description: The investigator's objective assessment of ocular health assessed for each study Pair after 3 days wear by biomicroscopy. Bulbar and Limbal Hyperemia; Corneal Staining Type, Extent and Depth, Conjunctival Staining and Indentation. BrienHolden Vision Institute Continuous Scale: 1-4, 0.5 steps (1=Very, 2=Slight, 3=Moderate, 4=Severe)
Time Frame: 3 Days Follow-up
Population: Only right eye data shown. Left eye data virtually identical. One subject had non-contact lens related adverse event in the nelfilcon A group. Subject temporarily discontinued and went on to complete the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Number analyzed (Participants) | 16 | 14 | 30
units on a scale
  Bulbar Hyperemia (Nasal) | 0.88 (0.2) | 0.96 (0.3) | 0.95 (0.4)
  Bulbar Hyperemia (Temporal) | 0.81 (0.3) | 0.96 (0.2) | 0.98 (0.4)
  Bulbar Hyperemia (Superior) | 0.63 (0.4) | 0.64 (0.5) | 0.72 (0.5)
  Bulbar Hyperemia (Inferior) | 0.72 (0.4) | 0.64 (0.5) | 0.75 (0.5)
  Limbal Hyperemia (Nasal) | 0.53 (0.5) | 0.96 (0.7) | 0.47 (0.6)
  Limbal Hyperemia (Temporal) | 0.44 (0.4) | 0.89 (0.7) | 0.38 (0.5)
  Limbal Hyperemia (Superior) | 0.38 (0.4) | 0.68 (0.7) | 0.30 (0.4)
  Limbal Hyperemia (Inferior) | 0.41 (0.5) | 0.75 (0.8) | 0.33 (0.5)
  Corneal Staining Type (Central) | 0.00 (0.0) | 0.18 (0.5) | 0.17 (0.6)
  Corneal Staining Type (Nasal) | 0.19 (0.8) | 0.14 (0.5) | 0.07 (0.4)
  Corneal Staining Type (Temporal) | 0.16 (0.4) | 0.25 (0.7) | 0.32 (0.8)
  Corneal Staining Type (Superior) | 0.34 (0.7) | 0.07 (0.3) | 0.38 (0.8)
  Corneal Staining Type (Inferior) | 0.50 (1.0) | 0.50 (0.9) | 0.67 (0.9)
  Corneal Staining Extent (Central) | 0.00 (0.0) | 0.07 (0.2) | 0.08 (0.3)
  Corneal Staining Extent (Nasal) | 0.03 (0.1) | 0.04 (0.1) | 0.02 (0.1)
  Corneal Staining Extent (Temporal) | 0.09 (0.3) | 0.11 (0.3) | 0.10 (0.2)
  Corneal Staining Extent (Superior) | 0.22 (0.4) | 0.04 (0.1) | 0.22 (0.5)
  Corneal Staining Extent (Inferior) | 0.41 (0.7) | 0.32 (0.6) | 0.38 (0.6)
  Corneal Staining Depth (Central) | 0.00 (0.0) | 0.14 (0.4) | 0.10 (0.3)
  Corneal Staining Depth (Nasal) | 0.06 (0.3) | 0.07 (0.3) | 0.03 (0.2)
  Corneal Staining Depth (Temporal) | 0.13 (0.3) | 0.14 (0.4) | 0.17 (0.4)
  Corneal Staining Depth (Superior) | .025 (0.5) | 0.07 (0.3) | 0.20 (0.4)
  Corneal Staining Depth (Inferior) | 0.25 (0.5) | 0.29 (0.5) | 0.40 (0.5)
  Conjunctival Staining (Nasal) | 0.34 (0.6) | 1.29 (1.2) | 1.65 (0.9)
  Conjunctival Staining (Temporal) | 0.28 (0.5) | 0.68 (0.9) | 1.65 (0.9)
  Conjunctival Staining (Superior) | 0.13 (0.3) | 0.04 (0.1) | 1.48 (0.8)
  Conjunctival Staining (Inferior) | 0.19 (0.4) | 0.64 (0.9) | 1.55 (0.8)
  Conjunctival Indent (Nasal) | 0.00 (0.0) | 0.00 (0.0) | 0.28 (0.5)
  Conjunctival Indent (Temporal) | 0.00 (0.0) | 0.00 (0.0) | 0.28 (0.5)
  Conjunctival Indent (Superior) | 0.06 (0.3) | 0.00 (0.0) | 0.22 (0.5)
  Conjunctival Indent (Inferior) | 0.06 (0.3) | 0.00 (0.0) | 0.20 (0.5)

ADVERSE EVENTS:
Time Frame: From dispense up to 3 days for each study lenses
Arm/Group | Nelfilcon A | Etafilcon A | Filcon II 3
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14 | 0/30
Other Adverse Events (participants affected / at risk) | 1/16 | 0/14 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nelfilcon A (N=16) | Etafilcon A (N=14) | Filcon II 3 (N=30)
Non-lens related (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — Only right eye data shown. Left eye data virtually identical. One subject had non-contact lens related adverse event in the nelfilcon A group. Subject temporarily discontinued and went on to complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor.